CLINICAL TRIAL: NCT05170984
Title: A Prospective Cohort Survey of Foot and Leg Chronic Wounds Followed up to 20 Weeks After Initiation of CACIPLIQ20® add-on to Optimal Local Care
Brief Title: MAtrix Therapy for Hard-to-heal ChrOnic Wounds
Acronym: MATHCOW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Organ, Tissue, Regeneration, Repair and Replacement (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-A01910-41
Record Dates: First submitted 2021-11-23; First posted 2021-12-28 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Chronic Ulcer of Leg or Foot; Diabetic Foot Ulcer; Arterial Ulcer; Venous Ulcer of Leg
Keywords: CACIPLIQ20; Chronic Wound; Chronic Ulcer; Hard-to-heal Wound
MeSH Terms: conditions — Diabetic Foot; Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CACIPLIQ20® (Experimental): Treatment of the target wound with CACIPLIQ20® in addition to optimal local care
  Interventions: Device: CACIPLIQ20®

INTERVENTIONS:
Device: CACIPLIQ20® — Application of CACIPLIQ20® by spray, directly on the wound surface, after wound cleaning and debridement, twice a week, until wound closure (or up to 20 weeks maximum).

SUMMARY:
CACIPLIQ20® is currently a class III CE marked medical device available in various European and non-European countries, and currently primarily used in managing hard-to-heal wounds.

This study is a prospective and standardized recording of patients' data followed in real-life conditions to appreciate the benefits of a therapeutic strategy including CACIPLIQ20® use. It also aims at collecting data to follow-up the device's efficacy and safety and estimate its cost-effectiveness.

DETAILED DESCRIPTION:
§ Study context:

CACIPLIQ20® is a bioengineered structural analogue of heparan sulfate glycosaminoglycans. Numerous experimental studies have provided strong evidence that CACIPLIQ20® promotes tissue regeneration by reconstructing the cellular microenvironment following tissue injury. Case studies collected in various clinical settings support the clinical interest of CACIPLIQ20® in the management of hard-to-heal chronic wounds.

CACIPLIQ20® is currently a class III CE marked medical device (NSAI-0050 CE MARK ECDEC-NL-A4) with the following indications:

Chronic ulcers showing no tendency to heal after 6 months of standard care, or still unhealed after 12 months, such as:

* Pressure ulcers;
* Peripheral arterial disease (such as Stage IV Leriche & Fontaine) ulcers;
* Diabetic ulcers (including amputation).

CACIPLIQ20® is available in various European and non-European countries and currently primarily used in managing hard-to-heal wounds.

Therefore, there is an opportunity to organize a prospective and standardized recording of patients' data followed in real-life conditions to appreciate the benefits of a therapeutic strategy including CACIPLIQ20® use and to collect data that may help to highlight its efficacy and safety and estimate its cost-effectiveness.

§ Hard-to-heal leg/foot ulcerations:

Leg ulcers of venous, mixed or arterial origin as well as neuropathic or neuroischaemic diabetic foot ulcers represent the most prevalent chronic wounds followed and managed in daily practices.

Arterial leg ulcers and Diabetic foot ulcers (DFU)s (especially for neuroischaemic DFUs) have frequently a rather poor healing prognosis despite revascularization attempts and application of best local cares including, for DFUs, wearing of appropriate off-loading devices. The risk of deciding minor or major lower limb amputation is high and the chance to obtain wound closure at 20-24 weeks is, at the best, around 20-30%.

For leg ulcers of venous origin (ankle brachial pressure index (ABPI) ≥0.8) or of mixed origin (ABPI ranges between 0.6 and 0.8), the healing prognosis is better with application of best local cares and the use when the ABPI is >0.7 or 0.8 of an efficient venous bandaging. Nevertheless, when initiating the management of large old wounds (area >10 cm² and ulcer present for at least 6 months) the chance to obtain wound closure at 20-24 weeks is of 20-30% at best.

This survey will specifically include patients presenting a hard-to-heal foot/leg ulceration such as: leg ulcers of predominantly venous origin but with an ulcer surface >10 cm² and/or an estimated wound duration of at least 5 months, leg ulcer with arterial participation including critical limb ischemia, or neuropathic and neuroischaemic DFUs.

§ Study organization:

The inclusion of patients is decided the day when the addition of CACIPLIQ20® to the standard of local care is decided. The follow-up of the patient in the cohort will be carried out until the target wound is closed or up to a maximum of 20 weeks.

The inclusion and follow-up of patients are ensured, in agreement and in cooperation with the healthcare team of the subject, by doctors and expert nurses from the Cicat Occitanie network. This network relies on secured and validated teleconsultation tools. The inclusion of a patient in the cohort will not change the usual functioning of the network.

ELIGIBILITY:
General Inclusion Criteria:

* Patients justifying a treatment with CACIPLIQ20® according to a care provider.
* Patients presenting with a chronic wound that has not shown signs of improvement following treatment for at least 6 months prior to inclusion into the study.
* Adult patients of either gender aged at least 18 and without upper limit for age.
* Patients having received a full written and oral information about study conduct and objectives and having given a written consent to participate according to local regulations.
* Patients being seen as outpatients and for whom no hospitalization is expected/planned in the 6 forthcoming weeks.
* Patients who can and are willing to be followed by a study investigator for the duration of the study.
* Patients benefiting from a valid health insurance or social security coverage.

Target Wound Inclusion Criteria:

* Current wound that has not been previously treated with CACIPLIQ20®.
* Target wound located below the knee.
* Target wound is either:

  1. a leg ulceration predominantly of venous origin (no ischemia as previously defined) with an area >10 cm² and/or a duration of at least 5 months,
  2. a leg ulceration of any size or duration, with a documented ischemic lower limb problem,
  3. a foot ulceration of any size or duration, documented as a diabetic foot ulceration (DFU).
* If more than one wound is present and eligible, investigators will be required to select one as the target wound for this study. This wound should be the largest one. If wounds are of similar size, the ulceration considered by the investigator as the worst will be selected.

Exclusion Criteria:

* Female patients who are pregnant, or lactating.
* Bedridden patients unable to spend at least one hour per day sitting in a chair.
* Patients suffering from severe cognitive problems precluding any voluntary participation to the study.
* Patients with, according to investigator's opinion, a very poor life expectancy.
* Patients with leg or foot ulcerations which are not of venous, arterial or diabetic origin (e.g. Martell's ulcer and related ulcers, pressure ulcers, traumatic wounds or burns)
* Patients whose target wound is located on an amputation stump.
* Patients presenting with a fungating wound at the time of inclusion.
* Patients in an emergency situation and unable to give consent.
* Patients intolerant to one of the study device components or to heparinoids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Rate of wound closure | Within 20 weeks after treatment initiation
  Wound closure defined as a 100% re-epithelialization, including:
  * A confirmed complete closure (CCC), defined as a wound closure notified by investigator and confirmed by an independent reviewer when analysing wound photos.
  * A possible complete closure (PCC), defined as a wound closure notified by investigator without confirmation by the independent reviewer (either no photo or photo of too poor quality or no unambiguous confirmation).
  The primary endpoint is the sum of CCC and PCC.

SECONDARY OUTCOMES:
Rate of adverse events (AEs) related to CACIPLIQ20® use | From baseline to wound closure or 20 weeks after treatment initiation
  Rate of adverse events (AEs) occurring during the study course including serious and non-serious AEs, anticipated or unanticipated AEs, related to CACIPLIQ20® use, according to investigators' opinion.
Rate of device deficiencies (DDs) | From baseline to wound closure or 20 weeks after treatment initiation
  Rate of device deficiencies (DDs) occurring during the study course including anticipated or unanticipated DDs.
Rate of wound closure according to the type of closure (CCC, PCC) and according to the nature of the treated wounds (Venous Leg Ulcers, Arterial Ulcers and Diabetic Foot Ulcers). | Within 20 weeks after treatment initiation
Time to wound closure | Within 20 weeks after treatment initiation
Changes in the Pain Visual Analogic Scale | From baseline to wound closure or 20 weeks after treatment initiation
  Pain Visual Analogic Scale from 0 (no pain) to 10 (unbearable pain)

CONTACTS AND LOCATIONS:
Overall Officials: Luc TEOT, MD, PhD, Principal Investigator — Réseau Cicat-Occitanie
Locations (1):
- Réseau Cicat-Occitanie, Montpellier, France

IPD SHARING:
Plan to Share IPD: No